CLINICAL TRIAL: NCT00950872
Title: A Prospective, Single-Center Investigation of the Safety and Performance of the ENDO GIA Staplers With ENDO GIA Single Use Loading Units With DUET TRS TM in a Gastric Bypass Procedure
Brief Title: Safety and Efficacy Study of Duet TRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AS08016
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-03

CONDITIONS: Roux En Y Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duet TRS (Experimental): Subjects receive Duet TRS
  Interventions: Device: Duet TRS

INTERVENTIONS:
Device: Duet TRS — Patients will have their gastric pouch created with ENDO GIA staplers with Single Use Loading Units with Duet TRS.

SUMMARY:
The objectives of this clinical trial are the overall performance and safety of the ENDO GIA Staplers with ENDO GIA SULUs with Duet TRS TM.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18-65 years of age.
* The patient has a BMI of 40-60 kg/m2 or 35-40 kg/m2 with comorbidities
* The patient must be willing and able to participate in the study procedures and able to understand and sign the informed consent.

Exclusion Criteria:

* The procedure is needed as revision bariatric surgery or the patient has had prior gastric surgery (nissen fundoplication, hiatal hernia, etc)
* The patient is pregnant.
* The patient has an active, or history of, infection at the operative site.
* The patient is unable or unwilling to comply with the study requirements, follow-up schedule, or to give valid informed consent.
* Patient has an abdominal ventral hernia
* The patient has a history of liver disease
* The patient has a history of drug or alcohol abuse
* The patient has a history of venous thrombosis or pulmonary embolism
* The patient has a history of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Pryor, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 24, 2009 and March 29, 2010, a total of 29 patients were consented and screened for potential study participation at one institution (Duke University). Of the 29 eligible patients, 2 did not have surgery resulting in a total of 27 patients for the analysis.
Pre-assignment Details: Subjects were evaluated for pre-operative and intra-operative eligibility criteria prior to enrollment.
Groups:
- Duet TRS: Duet TRS is a staple line buttress
Period: Overall Study
Arm/Group | Duet TRS
Started | 29
Completed | 26
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Did not have surgery | 2

BASELINE CHARACTERISTICS:
Population: number of subjects consented
Arm/Group | Duet TRS
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (11.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 17
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events.
Time Frame: Day 30
Population: Of the 29 eligible patients, 2 did not have surgery resulting in a total of 27 patients for the analysis.
Measure: Number; unit: adverse events
Arm/Group | Duet TRS
Number analyzed (Participants) | 27
adverse events | 6

2. Secondary Outcome: Operating Room (OR) Time
Description: OR time was captured in minutes, with time starting at the first port placement and concluding at the removal of the last port.
Time Frame: Day 0
Population: Of the 29 eligible patients, 2 did not have surgery resulting in a total of 27 patients for the analysis.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Duet TRS
Number analyzed (Participants) | 27
minutes | 98 (27) [62 to 165]

3. Secondary Outcome: Length of Hospital Stay
Description: Days spent in the hospital
Time Frame: Day 2 (Approximately 1.5 days post randomization)
Population: Of the 29 eligible patients, 2 did not have surgery resulting in a total of 27 patients for the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Duet TRS
Number analyzed (Participants) | 27
days | 1.5 (0.6) [1 to 3]

4. Secondary Outcome: Incidence of Stapler 'Misfires'
Description: The incidence of stapler misfires was captured as the number of patients with misfires. The types of misfires that were captured were less than B shaped staples, incomplete staple line and stripping of the rack teeth.
Time Frame: Day 0
Population: Of the 29 eligible patients, 2 did not have surgery resulting in a total of 27 patients for the analysis.
Measure: Number; unit: participants
Arm/Group | Duet TRS
Number analyzed (Participants) | 27
participants | 3

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Duet TRS
Serious Adverse Events (participants affected / at risk) | 2/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duet TRS (N=27)
Gastrojejunal Anatomosis Stricture (Gastrointestinal disorders) | 2 (2) — Of the 29 eligible patients, 2 did not have surgery resulting in a total of 27 patients for the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No